CLINICAL TRIAL: NCT03423836
Title: Maternal Oral Therapy to Reduce Obstetric Risk Kids
Acronym: MOTORKids
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 07-0727; 3U01DE014577-04S1 (NIH)
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Periodontitis; Autism; Premature Infants
MeSH Terms: conditions — Periodontitis; Autistic Disorder; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Risk Infants: Motor infants born prior to 35 weeks gestational age, or, infants small (<10th percentile) for gestational age.
- Low Risk Infants: Motor infants born after the completion of the 37th week of gestation and appropriate for gestational age.

SUMMARY:
The principal objective was to conduct a 5 year; multi-center, observational follow-up study enrolling infants born to mothers who participated in the MOTOR clinical trial to determine the effects of maternal periodontal therapy during pregnancy on neonatal morbidity and mortality and whether this will result in lower incidence of functional neurological impairment.

DETAILED DESCRIPTION:
A total of 525 infants where planned to be enrolled at the 3 performance sites. The number of infants enrolled at each site depended on past Motor recruitment rates, and the observed delivery rate of high risk babies at that site. Infants were enrolled from both the high risk and low risk groups. The intended sample size was fixed, over sampling among the low risk group and was used to assure the sample size.

The Data Coordinating Center (DCC) identified and provided each clinical site with participant listings of all MOTOR high risk births and a randomly ordered sample of low risk births for enrollment into the study.

Mothers where approached by MOTOR or MOTORkids personnel to ascertain participant interest in enrolling their infant. Once consent was obtained, infants were followed and tracked until scheduled for the follow-up exams at age 24 months +/- 2 months adjusted age.

ELIGIBILITY:
Inclusion Criteria:

* All infants born to mothers enrolled to MOTOR study prior to 35 weeks gestational age,
* All small for gestational age (SGA) infants and all infants born after 37 weeks gestation and who were appropriate for gestational age are eligible for enrollment.
* All infants born < 34 weeks gestation and all SGA infants will be considered a high risk infant and will be recruited for enrollment.
* Appropriate weight for gestational age infants born after 37 weeks will be considered low risk infants and a random sample of these infants will be recruited for enrollment.

Exclusion Criteria:

* Only a random sample of the low risk group will be recruited.

Min Age: 1 Day | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A total of 525 infants are planned to be enrolled at the 3 performance sites. The number of infants enrolled at each site will depend on their past Motor recruitment rates, and the observed delivery rate of high risk babies at that site. Infants will be enrolled from both the high risk and low risk group. This rate of enrollment is expected to vary by 10% to 20% across the sites. It is expected that sites will enroll 3-6 infants a month over a 3 year period. The intended sample size is fixed, over sampling among the low risk group will be used to assure the sample size.
Sampling Method: Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2007-04-30 (Actual); Primary Completion 2010-05-31 (Actual); Study Completion 2013-01-11 (Actual)

PRIMARY OUTCOMES:
MCHAT Score | 24 months
  MCHAT composite risk score for Autism questionnaire is a 20-item screening tool completed by parents of children aged 16-30 months to evaluate Autism Spectrum Disorder (ASD) risk. Score ranges include 0 to 20 with 2 or less indicating low-risk, 3-7 medium-risk and 8-20 indicating high-risk.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Bose, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (4):
- United States (4):
  - University of Alabama at Birmingham Department of Ostetrics and Gynecology, Birmingham, Alabama
  - Department of Periodontology, UNC School of Dentistry, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - University of Texas Health Science Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bose C, Valentine GC, Philips K, Boggess K, Moss K, Barros SP, Marchesan J, Wu D, O'Shea TM, Peralta-Carcelen M, Goldstein R, Ramamurthy R, Beck JD. Antepartum periodontitis treatment and risk of offspring screening positive for autism spectrum disorder. J Perinatol. 2023 Apr;43(4):470-476. doi: 10.1038/s41372-023-01610-x. Epub 2023 Jan 25. PMID 36697694